CLINICAL TRIAL: NCT03935334
Title: A Randomized, Multicenter, Double-blind Clinical Trial Comparing Pharmacodynamic, Pharmacokinetic and Safety of a Biosimilar Eptacog Alfa (AryoSeven) and Novoseven®, in Patients With Hemophilia A or B With Inhibitors.
Brief Title: Clinical Trial Comparing a Biosimilar Eptacog Alfa With Novoseven, in Patients With Hemophilia With Inhibitors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AryoGen Pharmed Co. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UGA 2014-01
Record Dates: First submitted 2019-04-29; First posted 2019-05-02 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2020-07

CONDITIONS: Hemophilia A or B With Inhibitor
MeSH Terms: conditions — Hemophilia A | interventions — recombinant FVIIa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding will be performed by an independent third party operator (nurse/pharmacist, unblinded), who will prepare undistinguishable syringes with patient's dosing and labelling.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eptacog alfa, biosimilar (AryoSeven) (Experimental): Patients will be randomized to receive, in a 2x2 crossover setting, either a single dose of biosimilar eptacog alfa, activated (AryoSeven) of 90 μg/kg or 270 μg/kg, or eptacog alfa, activated (Novoseven) of 90 μg/kg or 270 μg/kg, or vice-versa, separated by a washout period of 3 days.
  Interventions: Biological: Biosimilar eptacog alfa, activated (AryoSeven)
- Novoseven (Active Comparator): Patients will be randomized to receive, in a 2x2 crossover setting, either a single dose of biosimilar eptacog alfa, activated (AryoSeven) of 90 μg/kg or 270 μg/kg, or eptacog alfa, activated (Novoseven) of 90 μg/kg or 270 μg/kg, or vice-versa, separated by a washout period of 3 days.
  Interventions: Biological: Eptacog alfa, activated (Novoseven)

INTERVENTIONS:
Biological: Biosimilar eptacog alfa, activated (AryoSeven) — A single dose of eptacog alfa biosimilar (AryoSeven) 90 μg/kg or 270 μg/kg. Then, in an open follow up phase of 12 months, for every bleeding episode patients will receive eptacog alfa biosimilar, on demand, for one of more days until resolution of bleeding, based on the Investigator's decision - or - prophylaxis with eptacog alfa biosimilar, with dose, frequency, and duration of treatment based on the Investigator's decision. The modality of treatment (on demand or prophylaxis) will be decided by the Investigator.
  Arms: Eptacog alfa, biosimilar (AryoSeven)
Biological: Eptacog alfa, activated (Novoseven) — A single dose of eptacog alfa (Novoseven) 90 μg/kg or 270 μg/kg. Then, in an open follow up phase of 12 months, for every bleeding episode patients will receive eptacog alfa biosimilar, on demand, for one of more days until resolution of bleeding, based on the Investigator's decision - or - prophylaxis with eptacog alfa biosimilar, with dose, frequency, and duration of treatment based on the Investigator's decision. The modality of treatment (on demand or prophylaxis) will be decided by the Investigator.
  Arms: Novoseven

SUMMARY:
The purpose of this multicentre, randomized, double-blinded, single dose, two-way cross-over study, is to compare the pharmacokinetics (PK) and pharmacodynamic (PD) of two different doses of the biosimilar eptacog alfa (activated) with Novoseven in 48 patients, adult and children (>12 years), not bleeding, with hemophilia A or B with inhibitors. Patients will be randomized to receive either a single dose of eptacog alfa biosimilar 90 μg/kg or 270 μg/kg and one single dose of NovoSeven 90 μg/kg or 270 μg/kg, or vice versa, with doses separated by a washout period. All patients will be followed 12 months and will receive biosimilar eptacog alfa, on demand, for every bleeding episode that should occur - or - for prophylaxis, with the aim of monitoring of inhibiting antibody formation, lack of efficacy and collection of safety data.

DETAILED DESCRIPTION:
Forty-eight patients enrolled, not bleeding, will be randomized to receive two injections separated by a washout period of 3 days (t1/2 = 2.3h). Patients are centrally registered and randomized to receive in a 2x2 cross-over setting either a single dose of two for the following products: A: AryoSeven 90 µg/kg and B: NovoSeven 90 µg/kg - or - C: AryoSeven 270 µg/kg and D: NovoSeven 270 µg/kg.

Patients will be hospitalized at the time of study medication administration and plasma sampling. Before any treatment, a blood sample will be obtained in all patients for testing for immunogenicity.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of congenital hemophilia A or B with inhibitors to FVIII or FIX titer >5 Bethesda Units (BU)
* with > 2 episodes of bleeding/year requiring treatment with FVII infusions, non in bleeding status
* male subjects
* adult and children (>12 years)
* written informed consent to the protocol to be eligible for the study. For minor patients, parent/legal guardian will provide consent and, when possible, patient assent will also be obtained. For compromised patients, their designated proxy must provide informed consent.
* For the PK/PD phase, patients will be hospitalized at the time of study medication administration for plasma sampling (2 times during the study).

Exclusion Criteria:

* Any other type of congenital or acquired coagulopathy, such as liver disease (hepatitis), vitamin k deficiency, uremia, malignancy.
* Antibodies against Factor VII
* Ongoing bleeding prophylaxis regimens with Novoseven or planned to occur during the trial
* Patients who have received routine (prophylactic) treatment with rFVIIa in the period between screening visit (visit 1) and visit 2 of this study (first dose administration)
* Platelet count less than 100.000 platelets/microliter (at screening visit)
* Any clinical sign or known history of an arterial thrombotic event or deep venous- thrombosis or pulmonary embolism
* HIV positive with current CD4+ count of less than 200/µL
* Liver cirrhosis
* Factor VIII/IX immune tolerance induction regimen planned to occur during the trial
* Known hypersensitivity to the study medication
* Parallel participation in another experimental drug trial.
* Parallel participation in another marketed drug trial that may affect the primary endpoint of the study

Min Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-02-03 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration time curve from time 0 to infinity, based on the last observed concentration (AUCinf) | Ten minutes prior to dose administration and at 10 minutes, 20 minutes, 1 hour, 3 hours, 5 hours, 8 hours, 12 hours, 24 hours and 30 hours after AryoSeven and NovoSeven injection
  Measurement of plasma level of factor VII clotting activity (FVII:C) determined by commercial Staclot® VIIa-recombinant tissue factor assay (Diagnostics Stago, France).
Treatment response to Thrombin Generation Assay (TGA), D-Dimer, F1.2 prothrombin fragments. | Ten minutes prior to dose administration and at 10 minutes, 20 minutes, 1 hour, 3 hours, 5 hours, 8 hours, 12 hours, 24 hours and 30 hours after AryoSeven and NovoSeven injection
  Measurement of plasma levels based on standard methods recommended by the Subcommittee on the control of anticoagulation of the ISTH

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve from 0 to the last measurable time point (AUClast). | Ten minutes prior to dose administration and at 10 minutes, 20 minutes, 1 hour, 3 hours, 5 hours, 8 hours, 12 hours, 24 hours and 30 hours after AryoSeven and NovoSeven injection
  Measurement of plasma level of factor VII clotting activity (FVII:C) determined by commercial Staclot® VIIa-recombinant tissue factor assay
Maximum plasma concentration (Cmax) | Ten minutes prior to dose administration and at 10 minutes, 20 minutes, 1 hour, 3 hours, 5 hours, 8 hours, 12 hours, 24 hours and 30 hours after AryoSeven and NovoSeven injection
  Measurement of plasma level of factor VII clotting activity (FVII:C) determined by commercial Staclot® VIIa-recombinant tissue factor assay
Time of Cmax (tmax); | Ten minutes prior to dose administration and at 10 minutes, 20 minutes, 1 hour, 3 hours, 5 hours, 8 hours, 12 hours, 24 hours and 30 hours after AryoSeven and NovoSeven injection
  Measurement of plasma level of factor VII clotting activity (FVII:C) determined by commercial Staclot® VIIa-recombinant tissue factor assay
Fraction of the total AUCinf that was derived by extrapolation beyond tlast (AUCextra) | Ten minutes prior to dose administration and at 10 minutes, 20 minutes, 1 hour, 3 hours, 5 hours, 8 hours, 12 hours, 24 hours and 30 hours after AryoSeven and NovoSeven injection
  Measurement of plasma level of factor VII clotting activity (FVII:C) determined by commercial Staclot® VIIa-recombinant tissue factor assay
First order rate constant associated with the terminal (log-linear) portion of the curve (λz) | Ten minutes prior to dose administration and at 10 minutes, 20 minutes, 1 hour, 3 hours, 5 hours, 8 hours, 12 hours, 24 hours and 30 hours after AryoSeven and NovoSeven injection
  Measurement of plasma level of factor VII clotting activity (FVII:C) determined by commercial Staclot® VIIa-recombinant tissue factor assay
Elimination half-life | Ten minutes prior to dose administration and at 10 minutes, 20 minutes, 1 hour, 3 hours, 5 hours, 8 hours, 12 hours, 24 hours and 30 hours after AryoSeven and NovoSeven injection
  Measurement of plasma level of factor VII clotting activity (FVII:C) determined by commercial Staclot® VIIa-recombinant tissue factor assay
Mean residence time (MRT) | Ten minutes prior to dose administration and at 10 minutes, 20 minutes, 1 hour, 3 hours, 5 hours, 8 hours, 12 hours, 24 hours and 30 hours after AryoSeven and NovoSeven injection
  Measurement of plasma level of factor VII clotting activity (FVII:C) determined by commercial Staclot® VIIa-recombinant tissue factor assay
Clearance and CL/Dose (CL) | Ten minutes prior to dose administration and at 10 minutes, 20 minutes, 1 hour, 3 hours, 5 hours, 8 hours, 12 hours, 24 hours and 30 hours after AryoSeven and NovoSeven injection
  Measurement of plasma level of factor VII clotting activity (FVII:C) determined by commercial Staclot® VIIa-recombinant tissue factor assay
Volume of distribution (Vss) | Ten minutes prior to dose administration and at 10 minutes, 20 minutes, 1 hour, 3 hours, 5 hours, 8 hours, 12 hours, 24 hours and 30 hours after AryoSeven and NovoSeven injection
  Measurement of plasma level of factor VII clotting activity (FVII:C) determined by commercial Staclot® VIIa-recombinant tissue factor assay
Immunogenicity | On plasma samples obtained at screening visit, before the second dose/second drug administration, and then every 3 months for a year
  The Prothrombin Time (PT) based Bethesda assay will be used.
Adverse Events | Adverse events (AEs) will be monitored throughout the trial, from the first dose administered up to 12 months follow-up.
  Information about all adverse events, whether volunteered by the patient, discovered by investigator questioning, or detected through physical examination, laboratory test or other means, will be collected, recorded and followed as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Iacobelli, MD, Study Director — Consultant
Locations (8):
- Iran (3):
  - Hemophilia Center - Hematology & Oncology Dept. Shiraz University of Medical Science, Shiraz
  - Comprehensive Hemophilia Care Center, Tehran
  - Ali Asghar Hospital, Zahedan
- Turkey (Türkiye) (5):
  - Acibadem Adana Hastanesi, Pediatrik Hematoloji-Onkoloji Bölümü, Adana
  - Hacettepe Üniversitesi Çocuk Sağlığı ve Hastalıkları Anabilim Dalı Çocuk Hematolojisi Bilim Dalı, Ankara
  - Uludağ Üniversitesi Tıp Fakültesi Çocuk Sağlığı ve Hastalıkları Anabilim Dalı/Hematoloji Bilim Dalı, Bursa
  - Istanbul Üniversitesi Cerrahpaşa Tip Fakültesi Çocuk Sağlığı ve Hastalıkları Anabilim Dalı Çocuk Hematoloji-Onkoloji B.D., Istanbul
  - Ege Üniversitesi Tip Fakültesi Cocuk Sağliği ve Hastalikari Anabilim Dali ÇocukHematoloji Bilim Dali, Izmir

IPD SHARING:
Plan to Share IPD: No